CLINICAL TRIAL: NCT05981833
Title: A Randomized, Post-market Study Evaluating Dermal Allograft Augmentation of Large and Massive Rotator Cuff Tears
Brief Title: Dermal Allograft Augmentation of Large and Massive Rotator Cuff Tears
Status: Recruiting | Type: Observational
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AIRR-0094
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-03

CONDITIONS: Full-thickness Rotator Cuff Tear

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Repair without DAA: repaired without dermal allograft augmentation (DAA).
  Interventions: Device: Repair with DAA (dermal allograft augmentation)

INTERVENTIONS:
Device: Repair with DAA (dermal allograft augmentation) — Patients undergo rotator cuff repair with dermal allograft augmentation.

SUMMARY:
The purpose of this study is to compare postoperative healing of large and massive rotator cuff tears with preoperative MRI confirmed fatty infiltration stage II and higher repaired with or without dermal allograft augmentation (DAA).

DETAILED DESCRIPTION:
The primary objective is to evaluate postoperative healing of rotator cuff repair with and without DAA.

Primary: The primary outcome measure is healing evaluation in MRI . MRI Post-Operative Assessment (Goutallier Stage and Sugaya Classification)

Secondary: The secondary outcome measures are patient-reported outcome measures from validated outcome scoring systems, including:

American Shoulder and Elbow Surgeons Score (ASES)

Single Assessment Numeric Evaluation score (SANE)

Visual Analog Scale (VAS) for pain

Veterans RAND Health Survey (VR-12)

Population: Males and females between the ages of 30 and 75 years that require surgery for large and massive rotator cuff tears

Description of Treatment: Rotator cuff repair with or without augmentation using decellularized human dermal allograft.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between the ages of 30 and 75 years.
* Subject is planning to undergo arthroscopic surgery for full-thickness rotator cuff tear (RCT)
* Two complete RCTs or tear size equal to or greater than 3 cm in either the anterior-posterior or medial-lateral dimension
* Primary rotator cuff repair
* Stage II fatty infiltration or higher of the supraspinatus or infraspinatus muscle based on preoperative MRI6. Subject has a dual x-ray absorptiometry (DXA) or anterior posterior x-ray view of the target shoulder

Exclusion Criteria:

* The Subject is unable or unwilling to sign the patient informed consent, approved by the Institutional Review Board.
* The subject objects to the use of allograft
* Stage I or lower fatty infiltration of the supraspinatus AND infraspinatus muscle
* Complete full-thickness subscapularis tears of greater than the superior one third of the tendon (Lafosse grade 3 and above)
* Less than 2 mm joint space of the glenohumeral joint on either an anteroposterior or axillary radiograph
* Recurrent shoulder instability
* Corticosteroid injection in the operative shoulder within one month of surgery
* Revision rotator cuff repair
* Subject preoperative MRI obtained more than 12 months prior to surgery
* Pregnant or planning to become pregnant during the study period
* Workman's compensation case
* Subject has conditions or circumstances that would interfere with study requirements.

Intraoperative exclusion criteria:

Partial rotator cuff repairs

Lafosse grade 3 or higher subscapularis tears

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females between the ages of 30 and 75 years that require surgery for large and massive rotator cuff tears
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is healing evaluation in MRI | 26 Weeks
  MRI Post-Operative Assessment (Goutallier Stage and Sugaya Classification)
  MRI Post-Operative Assessment (Goutallier Stage and Sugaya Classification)

SECONDARY OUTCOMES:
The secondary outcome measures are patient-reported outcome measures from validated outcome scoring systems | Preop, 26 Weeks, 1 Year, 2 Year
  1. American Shoulder and Elbow Surgeons Score (ASES) A combination of objective measures and patient-reported outcomes, it measures pain and functional limitations in the shoulder. The objective questionnaire allows documentation of range of motion in the patient.
Single Assessment Numeric Evaluation score (SANE) | Preop, 26 Weeks, 1 Year, 2 Year
  Asks patients to rate shoulder pain as a percentage of normal.
Visual Analog Scale (VAS) for pain | Preop, two-week, six week, 26 Weeks, 1 Year, 2 Year
  The standard measure for pain on a 0-10 scale, 10 being the worst.
Veterans RAND Health Survey (VR-12) | Preop, 26 Weeks, 1 Year, 2 Year
  A self-administered health measure. Answers are summarized into two scores, a Physical Component Score and a Mental Component Score, which provides an important contrast between the respondents' physical and psychological health status.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Ruiz, MS, Study Director — Arthrex, Inc.
Locations (4):
- United States (4):
  - University of Arizona, Banner Health, Scottsdale, Arizona
  - Orthopaedic & Nuerosurgery Specialists, Greenwich, Connecticut
  - Southern Oregon Orthopedics Research Foundation, Medford, Oregon
  - Tennessee Orthopedic Foundation for Research Education and Research, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon J, Kim SH, Lee YH, Kim TI, Oh JH. The Rotator Cuff Healing Index: A New Scoring System to Predict Rotator Cuff Healing After Surgical Repair. Am J Sports Med. 2019 Jan;47(1):173-180. doi: 10.1177/0363546518810763. Epub 2018 Nov 28. PMID 30485753
- [Background] Duong JKH, Lam PH, Murrell GAC. Anteroposterior tear size, age, hospital, and case number are important predictors of repair integrity: an analysis of 1962 consecutive arthroscopic single-row rotator cuff repairs. J Shoulder Elbow Surg. 2021 Aug;30(8):1907-1914. doi: 10.1016/j.jse.2020.09.038. Epub 2020 Nov 4. PMID 33160028
- [Background] Pashuck TD, Hirahara AM, Cook JL, Cook CR, Andersen WJ, Smith MJ. Superior Capsular Reconstruction Using Dermal Allograft Is a Safe and Effective Treatment for Massive Irreparable Rotator Cuff Tears: 2-Year Clinical Outcomes. Arthroscopy. 2021 Feb;37(2):489-496.e1. doi: 10.1016/j.arthro.2020.10.014. Epub 2020 Oct 17. PMID 33080333
- [Background] Jackson GR, Bedi A, Denard PJ. Graft Augmentation of Repairable Rotator Cuff Tears: An Algorithmic Approach Based on Healing Rates. Arthroscopy. 2022 Jul;38(7):2342-2347. doi: 10.1016/j.arthro.2021.10.032. Epub 2021 Nov 10. PMID 34767956
- [Background] Omae H, Steinmann SP, Zhao C, Zobitz ME, Wongtriratanachai P, Sperling JW, An KN. Biomechanical effect of rotator cuff augmentation with an acellular dermal matrix graft: a cadaver study. Clin Biomech (Bristol). 2012 Oct;27(8):789-92. doi: 10.1016/j.clinbiomech.2012.05.001. Epub 2012 May 17. PMID 22607908
- [Background] Snyder SJ, Arnoczky SP, Bond JL, Dopirak R. Histologic evaluation of a biopsy specimen obtained 3 months after rotator cuff augmentation with GraftJacket Matrix. Arthroscopy. 2009 Mar;25(3):329-33. doi: 10.1016/j.arthro.2008.05.023. Epub 2008 Jul 24. PMID 19245998
- [Background] Barber FA, Burns JP, Deutsch A, Labbe MR, Litchfield RB. A prospective, randomized evaluation of acellular human dermal matrix augmentation for arthroscopic rotator cuff repair. Arthroscopy. 2012 Jan;28(1):8-15. doi: 10.1016/j.arthro.2011.06.038. Epub 2011 Oct 5. PMID 21978432
- [Background] Cummins CA, Murrell GA. Mode of failure for rotator cuff repair with suture anchors identified at revision surgery. J Shoulder Elbow Surg. 2003 Mar-Apr;12(2):128-33. doi: 10.1067/mse.2003.21. PMID 12700563
- [Background] Haque A, Pal Singh H. Does structural integrity following rotator cuff repair affect functional outcomes and pain scores? A meta-analysis. Shoulder Elbow. 2018 Jul;10(3):163-169. doi: 10.1177/1758573217731548. Epub 2017 Sep 25. PMID 29796103
- [Background] Sugaya H, Maeda K, Matsuki K, Moriishi J. Repair integrity and functional outcome after arthroscopic double-row rotator cuff repair. A prospective outcome study. J Bone Joint Surg Am. 2007 May;89(5):953-60. doi: 10.2106/JBJS.F.00512. PMID 17473131
- [Background] Mather J, MacDermid JC, Faber KJ, Athwal GS. Proximal humerus cortical bone thickness correlates with bone mineral density and can clinically rule out osteoporosis. J Shoulder Elbow Surg. 2013 Jun;22(6):732-8. doi: 10.1016/j.jse.2012.08.018. Epub 2012 Nov 22. PMID 23183030